CLINICAL TRIAL: NCT04522570
Title: Ultrasound Guided Percutaneous Thermal Ablation of Cervical Metastases From Thyroid Carcinoma
Brief Title: Thermal Ablation of Cervical Metastases From Thyroid Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1255/18
Record Dates: First submitted 2020-08-10; First posted 2020-08-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Neoplasia; Well-Differentiated Thyroid Cancer; Medullary Thyroid Cancer; Lymph Node Metastases
Keywords: differentiated thyroid cancer; medullary thyroid cancer; cervical lymph nodes; contrast-enhanced ultrasound; thermal ablation; laser ablation; radiofrequency ablation; cryoablation; elastography
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary; Lymphatic Metastasis | interventions — Laser Therapy; Cryosurgery; Cryoelectron Microscopy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- laser ablation (Active Comparator): Percutaneous Laser Ablation for the treatment of metastatic cervical lymph nodes with > 0.8 cm diameter with biopsy-proven diagnosis of differentiated thyroid carcinoma or medullary thyroid carcinoma.
  Interventions: Device: Laser ablation
- cryoablation (Active Comparator): Percutaneous cryoablation for the treatment of metastatic cervical lymph nodes with > 0.8 cm diameter with biopsy-proven diagnosis of differentiated thyroid carcinoma or medullary thyroid carcinoma.
  Interventions: Device: Cryoablation
- Radiofrequency ablation (Active Comparator): Percutaneous radio frequency ablation for the treatment of metastatic cervical lymph nodes with > 0.8 cm diameter with biopsy-proven diagnosis of differentiated thyroid carcinoma or medullary thyroid carcinoma.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Laser ablation — Single session with Diode laser ablation system; one or two applicators will be used for treatments; one to three illuminations; fixed output power of 3 watts (W); pullback technique; delivered energy: 1200-1800 Joules (J) varying according to tumor volume; treatment under local anesthesia +- conscious or moderate sedation;
  Other Names: LA
  Arms: laser ablation
Device: Cryoablation — Single session with Argon-based cryoablation system; one 17 Gauge (G) V-probe applicator will be used for treatments; fixed gas delivery of 100%; treatment under local anesthesia +- conscious or moderate sedation;
  Other Names: Cryo
  Arms: cryoablation
Device: Radiofrequency ablation — Single session with radiofrequency generator; one 17 Gauge (G) V-tip applicator with a 1 to 4cm active tip; moving-shot technique or multiple overlapping shot technique with 60 Watts (W) output power; treatment under local anesthesia +- conscious or moderate sedation;
  Other Names: RFA
  Arms: Radiofrequency ablation

SUMMARY:
This study will evaluate the clinical response and safety of ultrasound guided percutaneous thermal ablation of lymph node metastases from thyroid carcinoma as an alternative to surgical treatment.

The ablation of cervical lymph node metastases from differentiated thyroid carcinoma or medullary thyroid carcinoma will be directed to lesions larger than 0.8 cm, using ultrasound-guided radiofrequency ablation (RFA), laser ablation (LA) or cryoablation (Cryo) techniques, randomly assigned. Clinical and ultrasound monitoring will be carried out during 24 months, with examinations before the ablation procedure, immediately after including contrast-enhanced ultrasound (CEUS) when applicable, and B-mode, color Doppler and Shear-Wave elastography ultrasound follow up with 6, 12, and 24 months.

DETAILED DESCRIPTION:
Thyroidectomy is the main treatment of well differentiated thyroid carcinoma. Residual or recurrent cervical metastases are common (9-20% of patients during long-term follow up). Thermal ablation of cervical metastatic lymph nodes from thyroid carcinoma has been proposed in research centers as an option for the treatment of patients who remain with metastatic disease in cervical lymph nodes, despite thyroidectomy with or without neck dissection associated with radioiodine treatment. Potential advantages from percutaneous thermal ablation are related to less complication rates, less morbidity, possibility of outpatient treatment modality, and less global treatment costs when compared to the surgical approach.

Aims of the study:

1. To evaluate safety and efficacy of ultrasound-guided thermal ablation in the treatment of cervical lymph node metastases from differentiated thyroid carcinoma
2. To evaluate the best response to thermal ablation defined as lymph node reduction or volume stability after ablation
3. To evaluate the CEUS patterns of lymph nodes before and after ablation
4. To evaluate the elastography patterns of lymph nodes before and after ablation
5. To evaluate the tumor marker response after ablation
6. To evaluate the contribution of thermal ablation to decrease additional therapeutic procedures
7. To compare differences between LA, RFA and cryoablation in terms of complications, side effects and tolerability

Patients with cervical metastatic lymph nodes from differentiated thyroid carcinoma or medullary thyroid carcinoma who meet the eligibility criteria and who have been determined to be an appropriate candidate for local ablation therapy will be offered enrollment into the study. Patients agreeing to participate will become subjects of the study if they read and sign an informed consent form.

Treatment will be performed using three different ablation technologies (laser ablation, RFA or cryoablation) in a randomly assignment fashion.

Subjects will have up to six simultaneous treated lesions larger than 0.8 cm diameter with positive fine-needle aspiration biopsy. Ultrasound (and CEUS when applicable) will be performed over 24 months follow up in order to evaluate efficacy. Baseline and follow-up data will be collected for each subject via a web-based electronic data collection tool.

In case of recurrent disease treated by any ablative technique in patients who did not undergo previous neck dissection, a rescue neck dissection will be performed; in case of recurrent disease treated by any ablative technique in patients who underwent previous neck dissection, a new ablative technique approach will be considered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with fine needle aspiration biopsy (FNAb)-proven metastatic cervical lymph nodes at levels I, II, III, IV, V, VI or VII from differentiated thyroid carcinoma or medullary thyroid carcinoma who underwent total thyroidectomy and subsequent radioiodine therapy, in case of differentiated thyroid carcinoma.
* Patients considered high surgical risk candidate or patients who are informed about the ablation therapy and prefers it instead surgery;
* Patients with metastatic cervical lymph nodes over 0.8 cm diameter and under 4.0 cm diameter; no more than 6 simultaneous cervical nodal metastases;
* Cervical recurrences in previously lateral neck dissection patients for differentiated thyroid carcinoma or medullary thyroid carcinoma over 0.8 cm diameter.

Exclusion Criteria:

* Age under 18 years
* Uncorrectable coagulopathy;
* Inconclusive or benign cytologic specimens;
* Pregnancy or breast-feeding;
* Anaplastic or poor-differentiated thyroid carcinoma;
* Partial thyroidectomy
* Cervical tumors not considered to surgery (invading vessels, nerves, larynx or trachea);
* Serious medical illness, including any of the following: uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to the baseline visit, uncontrolled congestive heart failure;
* Participation in other studies that could affect the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of technical feasibility | immediately after the procedure
  defined as the ability to target the nodule and to perform ablation as preoperatively planned
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of thermal ablation of thyroid carcinoma cervical lymph node metastases | up to 4 weeks post-ablation
  Evaluation of minor and major complication rates, immediately after ablation; and one- and four-weeks post-ablation by telephone call.
  Minor and major complication rates [Designed as a safety issue: Yes]. The safety endpoint for this study is to assess the incidence and severity of procedure or device-related adverse events, as reported by the Common Terminology Criteria of Adverse Events - CTCAE V5. 2017 Version.

SECONDARY OUTCOMES:
Evaluation of technical success | immediately after the procedure
  Defined as the complete absence of color Doppler or, if applicable when tumors over 1.0 cm diameter, enhancement by contrast-enhanced ultrasound in the treated nodule
Evaluation of contrast-enhanced ultrasound pattern after thermal ablation therapy | 12 months
  Absence of enhancement is expected in treated cervical lymph nodes after local ablative therapy in comparison to pre-treatment enhancement pattern. Partial enhancement may indicate residual tumoral tissue requiring new ablation session
Evaluation of elastography pattern after thermal ablation therapy | 24 months
  Quantitative measurements of nodule stiffness designated by the most representative region of interest within the nodule estimating of Young's modulus in kilopascal (KPa) and shear wave velocity in centimetres per second (cm/s) of treated cervical lymph nodes after local ablative therapy in comparison to pre-treatment pattern.
Best response to the thermal ablation therapy | 24 months
  The best response is defined as a subject having local disease control related to lymph node volume reduction or volume stability in percentage will be assessed by ultrasound measurement in comparison to pre-treatment volume.
Evaluation of tumor marker response | 24 months
  Number of patients with tumor marker response: defined in negative thyroglobulin, calcitonin, or carcinoembryonic antigen (CEA) levels or anti-thyroglobulin antibodies
Evaluation of additional therapies | 24 months
  Number of patients with additional therapies: Additional therapies for persistent/recurrent local disease associated with the index tumor (s) under study or new cervical lymph node metastases.
Outcomes among thermal ablation therapies | 24 months
  Number of patients with complications, side effects and tolerability in each ablation technique.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo MC Freitas, PhD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within 18 months of study completion and for 6 months.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Hong YR, Luo ZY, Mo GQ, Wang P, Ye Q, Huang PT. Role of Contrast-Enhanced Ultrasound in the Pre-operative Diagnosis of Cervical Lymph Node Metastasis in Patients with Papillary Thyroid Carcinoma. Ultrasound Med Biol. 2017 Nov;43(11):2567-2575. doi: 10.1016/j.ultrasmedbio.2017.07.010. Epub 2017 Aug 12. PMID 28807450
- [Background] Guenette JP, Tuncali K, Himes N, Shyn PB, Lee TC. Percutaneous Image-Guided Cryoablation of Head and Neck Tumors for Local Control, Preservation of Functional Status, and Pain Relief. AJR Am J Roentgenol. 2017 Feb;208(2):453-458. doi: 10.2214/AJR.16.16446. Epub 2016 Nov 15. PMID 27845860
- [Background] Guang Y, Luo Y, Zhang Y, Zhang M, Li N, Zhang Y, Tang J. Efficacy and safety of percutaneous ultrasound guided radiofrequency ablation for treating cervical metastatic lymph nodes from papillary thyroid carcinoma. J Cancer Res Clin Oncol. 2017 Aug;143(8):1555-1562. doi: 10.1007/s00432-017-2386-6. Epub 2017 Mar 24. PMID 28342000
- [Background] Wang L, Ge M, Xu D, Chen L, Qian C, Shi K, Liu J, Chen Y. Ultrasonography-guided percutaneous radiofrequency ablation for cervical lymph node metastasis from thyroid carcinoma. J Cancer Res Ther. 2014 Nov;10 Suppl:C144-9. doi: 10.4103/0973-1482.145844. PMID 25450273
- [Background] Mauri G, Cova L, Ierace T, Baroli A, Di Mauro E, Pacella CM, Goldberg SN, Solbiati L. Treatment of Metastatic Lymph Nodes in the Neck from Papillary Thyroid Carcinoma with Percutaneous Laser Ablation. Cardiovasc Intervent Radiol. 2016 Jul;39(7):1023-30. doi: 10.1007/s00270-016-1313-6. Epub 2016 Feb 24. PMID 26911732
- [Background] Papini E, Bizzarri G, Bianchini A, Valle D, Misischi I, Guglielmi R, Salvatori M, Solbiati L, Crescenzi A, Pacella CM, Gharib H. Percutaneous ultrasound-guided laser ablation is effective for treating selected nodal metastases in papillary thyroid cancer. J Clin Endocrinol Metab. 2013 Jan;98(1):E92-7. doi: 10.1210/jc.2012-2991. Epub 2012 Nov 12. PMID 23150695
- [Background] Baudin E, Schlumberger M. New therapeutic approaches for metastatic thyroid carcinoma. Lancet Oncol. 2007 Feb;8(2):148-56. doi: 10.1016/S1470-2045(07)70034-7. PMID 17267329
- [Background] Monaco F. Classification of thyroid diseases: suggestions for a revision. J Clin Endocrinol Metab. 2003 Apr;88(4):1428-32. doi: 10.1210/jc.2002-021260. No abstract available. PMID 12679417
- [Background] Hegedus L. Clinical practice. The thyroid nodule. N Engl J Med. 2004 Oct 21;351(17):1764-71. doi: 10.1056/NEJMcp031436. No abstract available. PMID 15496625